CLINICAL TRIAL: NCT06328270
Title: Comparison of the Therapeutic Effects of Intra-Articular Injection of Ozone and Corticosteroid in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03.09.2019 / 2505
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The group received a 3-week intra-articular injection of 15 mg/ml ozone.
  Interventions: Other: Ozone - oxygen Therapy
- Control Group (Active Comparator): The group received a 1 ml intra-articular injection of betamethasone
  Interventions: Other: Corticosteroid

INTERVENTIONS:
Other: Ozone - oxygen Therapy — Ozone gas is a structurally unstable molecule that contains three oxygen atoms.
  Arms: Study Group
Other: Corticosteroid — 1 ml betamethasone
  Arms: Control Group

SUMMARY:
This clinical trial aimed to involve patients aged 40-85 years who had been experiencing knee pain for at least 6 months and had received a clinical diagnosis of knee osteoarthritis through radiologic imaging. The patients were randomly assigned to two groups. One group received a 3-week intra-articular injection of 15 mg/ml ozone, while the second group received a 1 ml intra-articular injection of betamethasone. All patients were evaluated before treatment, as well as 4 and 12 weeks after the first dose of treatment. The study evaluated treatment efficacy using the Visual Pain Score (VAS) and the Western Ontario and McMaster Universities Arthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

* 40-85 years old,
* have experienced knee pain and/or limited joint range of motion for at least 6 months,
* have a diagnosis of KOA supported by radiographic imaging.

Exclusion Criteria:

* patients had undergone knee joint surgery,
* had a history of previous intra-articular injections,
* had any rheumatological disease or malignancy,
* being pregnant,
* had pain radiating to the knee and leg.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Visual Pain Score | 4 weeks after the first dose of treatment
  Pain status of the patients was questioned with a scale between 0-10
Western Ontario and McMaster Universities Arthritis Index | 4 weeks after the first dose of treatment
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:[1] Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties

SECONDARY OUTCOMES:
Visual Pain Score | 12 weeks after the first dose of treatment
  Pain status of the patients was questioned with a scale between 0-10
Western Ontario and McMaster Universities Arthritis Index | 12 weeks after the first dose of treatment
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:[1] Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No